CLINICAL TRIAL: NCT01245322
Title: Extended Antimicrobial Treatment of Bacterial Vaginosis Combined With Human Lactobacilli to Find the Best Treatment and Minimize the Risk of Relapses
Brief Title: Treatment of Bacterial Vaginosis Combined With Human Lactobacilli
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skaraborg Hospital (Other Government)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Per-Goran Larsson, professor, Skaraborg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAV-3-BV
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Vaginosis
Keywords: treatment, lactobacilli
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactobacilli (Active Comparator): different lactobacilli.
  Interventions: Drug: lactobacilli

INTERVENTIONS:
Drug: lactobacilli — women were given a seven days course of daily 2% vaginal clindamycin cream (Dalacin vaginal cream 2%, Pfizer Norway Ltd) together with oral clindamycin 300 mg BID for 7 days (Dalacin 300 mg, Pfizer Norway Ltd). Oral clindamycin treatment was also given to the patient's sexual partner.
  Other Names: Treatments with differnt lactobacilli two zidovaltreatments

SUMMARY:
The primary objectives of this study were to characterize lactobacilli of human vaginal origin and to investigate if more extended antibiotic treatment against Bacterial Vaginosis, together with adjuvant lactobacilli treatment, could increase the cure rate and furthermore, to investigate factors that could influence relapse.

DETAILED DESCRIPTION:
Nine of the vaginal Lactobacillus strains isolated from healthy Swedish women and characterized in the present study were selected for the clinical trial.All women with symptomatic BV fulfilling the inclusion criteria were consecutively offered to participate in a prospective study of adjuvant lactobacilli given in addition to antibiotics. Women included were regularly menstruating women, 18 years or older, with normal gynaecological status, not pregnant or breast-feeding and without signs of other genital tract infections. Exclusion criteria were patients with hormonal intrauterine device without regular menstruation; women infected with Chlamydia trachomatis or with Trichomonas vaginalis, or with a clinical candida infection.

ELIGIBILITY:
Inclusion Criteria:

* were regularly menstruating women, 18 years or older, with normal gynaecological status, not pregnant or breast-feeding and without signs of other genital tract infections.

Exclusion Criteria:

* Exclusion criteria were patients with hormonal IUD without regular menstruation; women infected with Chlamydia trachomatis or with Trichomonas vaginalis, or with a clinical candida infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
characterize lactobacilli of human vaginal origin | 24 month
  characterize lactobacilli of human vaginal origin

SECONDARY OUTCOMES:
cure rate after 24 month | 24 month
  to investigate if more extended antibiotic treatment against BV, together with adjuvant lactobacilli treatment, could increase the cure rate and furthermore, to investigate factors that could influence relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Göran Larsson, professor, Principal Investigator — Skaraborg hospital and University College of Skövde, SE-541 85 Skövde, Sweden
Locations (1):
- Gynekologklinikken, Drammen, Norway

REFERENCES:
- [Derived] Larsson PG, Brandsborg E, Forsum U, Pendharkar S, Andersen KK, Nasic S, Hammarstrom L, Marcotte H. Extended antimicrobial treatment of bacterial vaginosis combined with human lactobacilli to find the best treatment and minimize the risk of relapses. BMC Infect Dis. 2011 Aug 19;11:223. doi: 10.1186/1471-2334-11-223. PMID 21854593